CLINICAL TRIAL: NCT04757649
Title: Suicide Prevention for Sexual and Gender Minority Youth (Case Series)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Aaron Blashill, Professor, San Diego State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HS-2020-0076 (1); 1R61MH120236-01 (NIH)
Record Dates: First submitted 2021-02-11; First posted 2021-02-17 (Actual); Results first posted 2023-05-03 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Suicide
Keywords: Sexual and gender minority youth; Patient Navigation; Safety Planning Intervention; Prevention
MeSH Terms: conditions — Suicide; Coitus

STUDY DESIGN:
Intervention Model Description: A broad recruitment strategy will be used to recruit participants within the greater San Diego. Potential participants will be requested to contact study personnel via email or telephone. A trained member of the study team will contact each potential participant to explain the study, obtain verbal consent for pre-enrollment screening, and conduct the screening process. For those who meet screening criteria, a trained member of the study team will provide more information about the study and engage in an informed consent process at an in-person appointment. Following informed consent, participants will complete self-report questionnaires and clinician-based interviews in person. At baseline and 3-month follow-up, participants will be asked to complete measures of suicidal coping and thwarted belongingness. At the 3-month follow-up, satisfaction with mental health services and satisfaction with interpersonal relationship with patient navigator will be assessed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Safety Planning Intervention with Navigation Services (Experimental): A patient navigation (PN) intervention for SGM youth/emerging adults designed to target mechanisms (i.e., decreasing thwarted belongingness and increasing suicide-related coping skills) that theoretically underlie suicide. The proposed intervention will integrate a single-session, empirically supported, suicide prevention intervention (Safety Planning Intervention; SPI) with PN services (PN+SPI). The patient navigator will deliver the SPI and continue frequent contact for the purpose of providing motivational enhancement, problem-solving, reinforcing coping strategies, and connecting participants to social support and mental health resources (e.g., SGM-specific support groups within the community).
  Interventions: Behavioral: Safety Planning Intervention with Navigation Services

INTERVENTIONS:
Behavioral: Safety Planning Intervention with Navigation Services — A patient navigation (PN) intervention for SGM youth/emerging adults designed to target mechanisms (i.e., decreasing thwarted belongingness and increasing suicide-related coping skills) that theoretically underlie suicide. The proposed intervention will integrate a single-session, empirically supported, suicide prevention intervention (Safety Planning Intervention; SPI) with PN services (PN+SPI). The patient navigator will deliver the SPI and continue frequent contact for the purpose of providing motivational enhancement, problem-solving, reinforcing coping strategies, and connecting participants to social support and mental health resources (e.g., SGM-specific support groups within the community).
  Other Names: PN+SPI Intervention

SUMMARY:
The overarching goal of this study is to develop a suicide prevention program for sexual-and-gender-minority youth and emerging adults. After development of the intervention program, a case series trial will be conducted to test the feasibility and acceptability of the intervention and study methods.

DETAILED DESCRIPTION:
Suicide is the 10th leading cause of death among all U.S. citizens, and is the 2nd leading cause of death among youth and emerging adults between the ages of 15 and 34. Moreover, U.S. representative data indicate increasing trends in suicide attempts and death by suicide. In addition to the immense psychological burden experienced by the family and friends of individuals who attempt and complete suicide, the costs of death by suicide and suicide attempts in 2013 were estimated at $93.5 billion.

One group that is particularly vulnerable to suicide is sexual and gender minorities (SGMs). SGM is an umbrella term used to describe individuals who identify as non-exclusively heterosexual (e.g., gay, lesbian, bisexual) and/or as transgender/non-binary (e.g., identify as a gender different from their birth sex). Extant research consistently notes substantial mental health disparities among SGMs in comparison to their heterosexual and cis-gender counterparts. In 2017, in the U.S., 23% of sexual minority youth reported one or more suicide attempts (in the past 12 months) vs. 5.4% of heterosexual youth. This disparity has also been noted in a meta-analysis of population-based longitudinal studies, with sexual minority adolescents and emerging adults reporting 2.26 increased odds of suicide attempts compared to their heterosexual counterparts. Prevalence of lifetime suicide attempts among gender minorities is also substantially elevated compared to the general population, with 45% of 18-24-year-old transgender individuals reporting history of one or more suicide attempts.

Despite these substantial health disparities in suicide among SGM youth/emerging adults, no known suicide prevention programs exist for this highly vulnerable population. Given this crucial gap in the literature, the proposed study will adapt and test a patient navigation (PN) intervention for SGM youth/emerging adults designed to target mechanisms (i.e., decreasing thwarted belongingness and increasing suicide-related coping skills) that theoretically underlie suicide. The proposed intervention will integrate a single-session, empirically supported, suicide prevention intervention (Safety Planning Intervention; SPI) with PN services (PN+SPI). The patient navigator will deliver the SPI and continue frequent contact for the purpose of providing motivational enhancement, problem-solving, reinforcing coping strategies, and connecting participants to social support and mental health resources (e.g., SGM-specific support groups within the community). This study will accomplish the following specific aims:

Specific Aim 1: To adapt and test an integrated PN+SPI designed to reduce suicide attempts among SGM youth and emerging adults. In this case series trial (N = 9), feasibility and acceptability of the PN+ SPI intervention will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age 15 to 29 years
* Identifies as gay, lesbian, bisexual, transgender, genderqueer, asexual, pansexual, non-binary, or another non-exclusively heterosexual identity, and/or reports same-gender romantic attraction, and/or reports same-gender sexual behavior in the past 12 months
* Resides in San Diego County, California
* Speaks English
* Is willing and able to provide informed consent
* Reports suicidal ideation over the past two weeks, as indicated by the clinician-administered Columbia-Suicide Severity Rating Scale (C-SSRS) Baseline version
* Reports a lifetime history of one or more suicide attempts

Exclusion Criteria:

* Individuals with immediate intention to attempt suicide will be excluded.

Ages: 15 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Identify as gay, lesbian, bisexual, transgender, genderqueer, asexual, pansexual, non-binary, or another non-exclusively heterosexual identity, and/or reports same-gender romantic attraction, and/or reports same-gender sexual behavior in the past 12 months.
Enrollment: 9 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron J Blashill, Principal Investigator — San Diego State University; Kristen J Wells, Principal Investigator — San Diego State University
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olfson M, Blanco C, Wall M, Liu SM, Saha TD, Pickering RP, Grant BF. National Trends in Suicide Attempts Among Adults in the United States. JAMA Psychiatry. 2017 Nov 1;74(11):1095-1103. doi: 10.1001/jamapsychiatry.2017.2582. PMID 28903161
- [Background] Ivey-Stephenson AZ, Crosby AE, Jack SPD, Haileyesus T, Kresnow-Sedacca MJ. Suicide Trends Among and Within Urbanization Levels by Sex, Race/Ethnicity, Age Group, and Mechanism of Death - United States, 2001-2015. MMWR Surveill Summ. 2017 Oct 6;66(18):1-16. doi: 10.15585/mmwr.ss6618a1. PMID 28981481
- [Background] Shepard DS, Gurewich D, Lwin AK, Reed GA Jr, Silverman MM. Suicide and Suicidal Attempts in the United States: Costs and Policy Implications. Suicide Life Threat Behav. 2016 Jun;46(3):352-62. doi: 10.1111/sltb.12225. Epub 2015 Oct 29. PMID 26511788
- [Background] Institute of Medicine (US) Committee on Lesbian, Gay, Bisexual, and Transgender Health Issues and Research Gaps and Opportunities. The Health of Lesbian, Gay, Bisexual, and Transgender People: Building a Foundation for Better Understanding. Washington (DC): National Academies Press (US); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK64806/ PMID 22013611
- [Background] Kann L, McManus T, Harris WA, Shanklin SL, Flint KH, Queen B, Lowry R, Chyen D, Whittle L, Thornton J, Lim C, Bradford D, Yamakawa Y, Leon M, Brener N, Ethier KA. Youth Risk Behavior Surveillance - United States, 2017. MMWR Surveill Summ. 2018 Jun 15;67(8):1-114. doi: 10.15585/mmwr.ss6708a1. PMID 29902162
- [Background] Miranda-Mendizabal A, Castellvi P, Pares-Badell O, Almenara J, Alonso I, Blasco MJ, Cebria A, Gabilondo A, Gili M, Lagares C, Piqueras JA, Roca M, Rodriguez-Marin J, Rodriguez-Jimenez T, Soto-Sanz V, Vilagut G, Alonso J. Sexual orientation and suicidal behaviour in adolescents and young adults: systematic review and meta-analysis. Br J Psychiatry. 2017 Aug;211(2):77-87. doi: 10.1192/bjp.bp.116.196345. Epub 2017 Mar 2. PMID 28254960
- [Background] Stanley B, Brown GK, Brenner LA, Galfalvy HC, Currier GW, Knox KL, Chaudhury SR, Bush AL, Green KL. Comparison of the Safety Planning Intervention With Follow-up vs Usual Care of Suicidal Patients Treated in the Emergency Department. JAMA Psychiatry. 2018 Sep 1;75(9):894-900. doi: 10.1001/jamapsychiatry.2018.1776. PMID 29998307
- [Background] Labouliere CD, Stanley B, Lake AM, Gould MS. Safety Planning on Crisis Lines: Feasibility, Acceptability, and Perceived Helpfulness of a Brief Intervention to Mitigate Future Suicide Risk. Suicide Life Threat Behav. 2020 Feb;50(1):29-41. doi: 10.1111/sltb.12554. Epub 2019 May 21. PMID 31112330
- [Background] Cramer RJ, Kapusta ND. A Social-Ecological Framework of Theory, Assessment, and Prevention of Suicide. Front Psychol. 2017 Oct 9;8:1756. doi: 10.3389/fpsyg.2017.01756. eCollection 2017. PMID 29062296
- [Derived] van der Star A, Randall A, Salgin L, Brady JP, Albright C, Mitzner J, Alexander J, Williams K, Weersing VR, Calzo JP, Rojas SA, Ramers CB, Wells KJ, Blashill AJ. Development of a Suicide Prevention Intervention for Sexual and Gender Minority Youth and Young Adults: Rationale, Design, and Evidence of Feasibility and Acceptability. Suicide Life Threat Behav. 2025 Apr;55(2):e70014. doi: 10.1111/sltb.70014. PMID 40179218

RESULTS

PARTICIPANT FLOW:
Recruitment Details: May 2021 through July 2021; San Diego County.
Period: Overall Study
Arm/Group | Safety Planning Intervention With Navigation Services
Started | 9
Completed | 7
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Safety Planning Intervention With Navigation Services
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 7
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender Identity: Male | 2
  Gender Identity: Female | 2
  Gender Identity: Trans Man | 1
  Gender Identity: Trans Woman | 1
  Gender Identity: Non-Binary | 1
  Gender Identity: Genderqueer | 1
  Gender Identity: Gender Non-Conforming | 0
  Gender Identity: Gender Fluid | 1
  Gender Identity: Agender | 0
  Gender Identity: Other Gender | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 1
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 9
Sexual Orientation [Count of Participants; unit: Participants]
  Gay/Lesbian | 3
  Bisexual | 5
  Straight/Heterosexual | 0
  Pansexual | 1
  Asexual | 0
  Questioning/I don't know | 0
  Other Sexual Orientation | 0

OUTCOME MEASURES:

1. Primary Outcome: The Interpersonal Needs Questionnaire-15 (INQ-15) - Thwarted Belongingness
Description: Assess thwarted belongingness (9 items on 7-point scales; scores range from 9 to 63 with higher scores indicating greater thwarted belongingness)
Time Frame: Cohen's d effect size as change from baseline thwarted belongingness scores at 3 months (0.00-0.49 small effect; 0.50-0.79 medium effect; 0.80-1.00 large effect)
Measure: Mean (95% Confidence Interval); unit: Cohen's d effect size
Arm/Group | Safety Planning Intervention With Navigation Services
Number analyzed (Participants) | 7
Cohen's d effect size | -0.29 [-1.42 to 0.85]

2. Primary Outcome: Suicide-Related Coping Scale (SRCS) - Internal Coping Skills
Description: Assess suicide-related internal coping skills (7 items on 5-point scales; scores range from 0 to 28 with higher scores indicating better internal coping)
Time Frame: Cohen's d effect size as change from baseline suicide-related internal coping scores at 3 months (0.00-0.49 small effect; 0.50-0.79 medium effect; 0.80-1.00 large effect)
Measure: Mean (95% Confidence Interval); unit: Cohen's d effect size
Arm/Group | Safety Planning Intervention With Navigation Services
Number analyzed (Participants) | 7
Cohen's d effect size | 0.67 [-0.50 to 1.83]

3. Primary Outcome: Suicide-Related Coping Scale (SRCS) - External Coping Skills
Description: Assess suicide-related external coping skills (7 items on 5-point scales; scores range from 0 to 28 with higher scores indicating better external coping)
Time Frame: Cohen's d effect size as change from baseline suicide-related external coping scores at 3 months (0.00-0.49 small effect; 0.50-0.79 medium effect; 0.80-1.00 large effect)
Measure: Mean (95% Confidence Interval); unit: Cohen's d effect size
Arm/Group | Safety Planning Intervention With Navigation Services
Number analyzed (Participants) | 7
Cohen's d effect size | 0.86 [-0.32 to 2.05]

ADVERSE EVENTS:
Time Frame: Three months
Description: An adverse event is defined as any untoward or unfavorable medical occurrence in a human participant, including any abnormal sign, symptom, or disease, temporally associated with participant's study participation, whether or not considered related to participant's study participation; it encompasses both physical and psychological harm. This study also included non-medical events that may be behavioral (i.e., self-harm) or social (e.g., child protective services involvement with the family).
Arm/Group | Safety Planning Intervention With Navigation Services
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 2/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Planning Intervention With Navigation Services (N=9)
Distress with increased suicidal ideation and emergency services involvement (Psychiatric disorders) | 1 (1) — Following arrest for misdemeanor, subject experienced distress and increased suicidal ideation, but they were able to engage safety plan and connect with mental health provider who contacted the Psychiatric Emergency Response Team.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Planning Intervention With Navigation Services (N=9)
Increased Anxiety (Psychiatric disorders) | 1 (1) — The content has been making the subject feel anxious outside of the study.
Arrest (Social circumstances) | 1 (1) — Subject was arrested for misdemeanor.

LIMITATIONS AND CAVEATS:
The study was conducted to assess the feasibility and acceptability of a newly developed suicide prevention intervention. By design, the quantitative outcome measurement was not sufficiently powered to evaluate preliminary efficacy and/or mechanistic target engagement.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT04757649/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT04757649/ICF_001.pdf